CLINICAL TRIAL: NCT05126550
Title: The Immunogenicity, Safety, and Effectiveness of the SARS-CoV-2 Vaccine (Vero Cell) Inactivated in Adult Population Aged 18 Years Old and Above in Indonesia
Brief Title: The Immunogenicity, Safety, and Effectiveness of the COVID-19 Inactivated Vaccine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PT. Kimia Farma (Persero) Tbk (Industry)
Responsible Party: Principal Investigator, Prenali Dwisthi Sattwika, Principal Investigator, Internist, Gadjah Mada University
Other Study IDs: Sinopharm21
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunogenicity: Group 1 constitutes the immunogenicity group which will be evaluated regarding immunogenicity, safety, and effectiveness of the SARS-CoV-2 vaccine (Vero cell) inactivated produced by Sinopharm
  Interventions: Biological: SARS-CoV-2 vaccine (Vero cell) inactivated
- Non-Immunogenicity: Group 2 that constitutes the non-immunogenicity group which will be evaluated regarding only safety and effectiveness of the aforementioned vaccine
  Interventions: Biological: SARS-CoV-2 vaccine (Vero cell) inactivated

INTERVENTIONS:
Biological: SARS-CoV-2 vaccine (Vero cell) inactivated — Two doses of 0.5 mL intramuscular injection containing 4 mcg (6.5 Unit) antigens with an interval of 21-28 days in accordance with "Vaksinasi Gotong Royong" (mutual cooperation vaccination program)

SUMMARY:
To fast respond the coronavirus disease of 2019 (COVID-19) pandemic, the Indonesian government has launched "Vaksinasi Gotong Royong" (a mutual cooperation vaccination program) in which any company/legal entity/business entity may purchase vaccines to be given free of charge to their employees and families of employees (The Indonesian Ministry of Health, 2021). Vaccines provided for this program include the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) inactivated vaccines produced by Sinopharm.

The Indonesian National Agency of Drug and Food Control (NADFC) has issued an Emergency Use Authorization (EUA) for several COVID-19 vaccines, including the SARS-CoV-2 vaccine (Vero cell) inactivated produced by Sinopharm (NADFC, 2021). Following EUA, Kimia Farma Indonesia as the holder of EUA has the obligation to monitor the safety and effectiveness in Indonesian population.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects aged 18 years old and above; Will receive the SARS-CoV-2 vaccine (Vero cell) inactivated produced by Sinopharm; Obtain informed consent to participate this study

Exclusion Criteria:

Previous SARS-CoV-2 vaccination, except for drop out after the first vaccine dose of more than 6 months ago; History of SARS-CoV-2 infection within the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruitment will target potential participants via local company/legal entity/business entity registering for "Vaksinasi Gotong Royong"
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-11-13 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The percent inhibition of SARS-CoV-2 surrogate Virus Neutralization Test neutralizing antibody (sVNT NAb) | At 14 days, 3 months, and 6 months after 2 doses of vaccination
  To evaluate the percent inhibition of SARS-CoV-2 sVNT NAb following the SARS-CoV-2 vaccine (Vero cell) inactivated administration at 14 days, 3 months, and 6 months after 2 doses of vaccination

SECONDARY OUTCOMES:
The geometric mean titer (GMT) of anti-spike protein receptor binding domain (sRBD) immunoglobulin G (IgG) antibody and the proportion of seropositivity of anti-nucleocapsid antibody | At 14 days, 3 months, and 6 months after 2 doses of vaccination
  To evaluate the GMT of anti-sRBD IgG antibody and the proportion of seropositivity of anti-nucleocapsid antibody following the SARS-CoV-2 vaccine (Vero cell) inactivated administration at 14 days, 3 months, and 6 months after 2 doses of vaccination
The proportion of adverse event following immunization | Within 28 days after 2 doses of vaccination
  To evaluate the proportion of adverse event following immunization (AEFI) following the SARS-CoV-2 vaccine (Vero cell) inactivated administration after the first dose until 28 days after the second dose of vaccination
The proportion of serious adverse event | Within 6 months after 2 doses of vaccination
  To evaluate the proportion of serious adverse event following the SARS-CoV-2 vaccine (Vero cell) inactivated administration after the first dose until 6 months after the second dose of vaccination
The proportion of symptomatic and PCR-confirmed SARS-CoV-2 infection | Within 6 months after 2 doses of vaccination
  To evaluate the proportion of symptomatic and PCR-confirmed SARS-CoV-2 infection following the SARS-CoV-2 vaccine (Vero cell) inactivated administration within 6 months after second dose of vaccination

CONTACTS AND LOCATIONS:
Locations (4):
- Indonesia (4):
  - Laboratorium Klinik Kimia Farma Diponegoro Bandung, Bandung
  - Laboratorium Klinik Kimia Farma Cikini, Jakarta
  - Laboratorium Klinik Kimia Farma Medan, Medan
  - Laboratorium Klinik Kimia Farma Sutomo Semarang, Semarang

IPD SHARING:
Plan to Share IPD: No